CLINICAL TRIAL: NCT04730011
Title: Short and Intensive Treatment of Children and Adolescents With Obsessive-Compulsive Disorder - A Study to Evaluate the Effectiveness of an Intensive Treatment Week: "A Future Without Constraint"
Brief Title: Short and Intensive Treatment of Children and Adolescents With Obsessive-Compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Susanne Walitza (Other)
Responsible Party: Sponsor-Investigator, Susanne Walitza, Head of the Department of Child and Adolescent Psychiatry, Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KJPP 2020-02053
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Patients are treated based on the Cognitive Behavioral Psychotherapy. This includes individual and group sessions over one week.
  Interventions: Behavioral: Short and Intensive Treatment

INTERVENTIONS:
Behavioral: Short and Intensive Treatment — Intensive Treatment Week with behavioural psychotherapy

SUMMARY:
Obsessive-compulsive disorders are very damaging illnesses; they can already appear in childhood and adolescence and become extremely chronic. With an average prevalence from 1-3%, they are among the most common psychiatric disorders in children and adolescents. 40% of diagnosed children and young adults display persistent and increasingly chronic symptoms and O-C disorders are highly complex syndromes with broadly varying manifestations. They arise from obsessive thoughts (ideas/thoughts or impulses, often senseless or tortured, that impose themselves or intrude) and obsessive behavior (ritualized patterns that must be frequently repeated).

ELIGIBILITY:
Inclusion Criteria:

* Obsessive-Compulsive Disorder diagnosis
* Male and female patients from 8-18 years
* Good German language speaking skills
* IQ of at least 75
* At least four days' participation in the treatment/therapy week
* Written agreement after clear explanation

Exclusion Criteria:

- No complete participation in the intensive week treatment/therapy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms severity of obsessive and compulsive symptoms in children and adolescents | 12 months
  The clinician-report questionnaire (BY-BOCS) contains 19 items designed to assess severity of obsessive and compulsive symptoms in children and adolescents.The test uses a 4-point scale to rate the severity of their obsessive compulsive behaviors. Higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Walitza, Prof. Dr. med. Dipl.-Psych., Principal Investigator — Sponsor GmbH
Locations (1):
- Psychiatric University Clinics, Department of Child and Adolescent Psychiatry, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No